CLINICAL TRIAL: NCT00186849
Title: Therapy for Children With Advanced Stage High Risk Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Wayne L. Furman, MD / Principal Investigator, St. Jude Children's Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NB-97
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2009-05-20 (Estimated); Status verified 2009-05

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Topotecan; Cyclophosphamide; Cisplatin; Doxorubicin; Etoposide; Ifosfamide; Carboplatin; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Drug: Topotecan, Cyclophosphamide, Cisplatin, Doxorubicin, Etoposide, Ifosfamide, Carboplatin; Procedure: Peripheral Blood Stem Cell Transplant

INTERVENTIONS:
Drug: Topotecan, Cyclophosphamide, Cisplatin, Doxorubicin, Etoposide, Ifosfamide, Carboplatin — See Detailed Description section for details of treatment interventions.
Procedure: Peripheral Blood Stem Cell Transplant — See Detailed Description section for details of treatment interventions.

SUMMARY:
This is a Phase II pilot study of chemotherapy and surgery for children with advanced stage high-risk neuroblastoma utilizing topotecan during an upfront window and other active agents during induction and intensification phases. The primary purpose is to estimate the response rate to an upfront window of two cycles of intravenous topotecan. We hypothesize that the topotecan window will be an effective therapy in terms of the response rate.

DETAILED DESCRIPTION:
In this prospective phase II trial, topotecan is administered intravenously daily for 5 days for each of 2 consecutive weeks for two cycles in an upfront treatment window. Patients subsequently will receive standard treatment during induction and intensification phases.

The objectives of this trial are:

* To estimate the response rate to an upfront window of two cycles of IV topotecan when given in doses adjusted to attain a targeted systemic exposure in children with advanced stage neuroblastoma.
* To determine the feasibility and toxicity of an intensification phase of high-dose chemotherapy with topotecan and cyclophosphamide followed by autologous peripheral blood stem cell transplant
* To estimate the 3-year overall survival and progression-free survival in patients treated with this approach
* To characterize the phenotype of neuroblastoma tumor cells
* To evaluate the disposition of topotecan in previously untreated patients with neuroblastoma

Details for chemotherapy intervention:

Window Phase Topotecan description, window therapy-Topotecan given intravenously daily as a 30 minute infusion for five consecutive days, off two days, and then five consecutive days. The dose for day 1 and 2 was 3.0 mg/m2 and subsequent doses were adjusted to attain a target systemic exposure. A second course of Topotecan was given approximately 16 days from the end of the first cycle, with the initial dose for the second course of Topotecan based on the dose required in the preceding course to attain the target AUC.

Induction Phase

Cyclophosphamide, MESNA, Adriamycin, Cisplatin, Carboplatin, and Etoposide description, Induction Phase (after completion of window) consists of 4 cycles of therapy:

Cycle 1:Cyclophosphamide 1 gm/m2 daily x 2 I.V. day 1 and 2 Adriamycin 35 mg/m2 I.V. day 1 only, MESNA: 250 mg/m2 I.V. immediately following cyclophosphamide infusion and at 3 and 6 hours post-infusion, and Etoposide: 30 mg/m2 over 30 minutes, followed by 250 mg/m2/day x 3 days I.V. by continuous infusion (days 2-5) Cycles 2 and 4- Cisplatin 40 mg/m2/day x 5 I.V. over 1 hour (days 1-5) Etoposide 200 mg/m2/day x 3 I.V. over 1 hour (days 2,3,4) Cycle 3: Carboplatin: dose adapted from GFR on day 1. Dose in mg/m2 = 8 x [(0.93 GFR) + 15] Ifosfamide: 2 gm/m2 I.V. over 1 hour daily x 3 (days 2, 3, 4) MESNA: 500 mg/m2 I.V. immediately after ifosfamide and 3 and 6 hours later Etoposide: 100 mg/m2 IV daily x 3 over 1 hour (days 2, 3, 4).

Intensification Phase

Topotecan, Cyclophosphamide, and MESNA- Intensification Therapy:

Topotecan - targeted dose - daily x 5 days for two weeks. Cyclophosphamide 750 mg/m2 IV over 1 hour on days 8 through 12. MESNA 175 mg/m2 IV immediately after cyclophosphamide and 3 and 6 hours later. Infusion of previously collected peripheral blood stem cells on day 14.

Subjects that do not respond to the Topotecan window will not receive topotecan during intensification, but instead will receive the following intensification therapy:

Carboplatin 700 mg/m2/day IV, over one hour q.o.d. x 3 Etoposide 500 mg/m2/day IV, over 6 hours q.o.d. x 3. Infusion of previously collected peripheral blood stem cells on day 8

Details for Intervention: Procedure/Surgery: Surgery Surgical resection will be performed after the window therapy in feasible subjects. If surgery was not possible after the Topotecan window resection of the primary tumor mass and careful lymph node staging was done after recovery from induction and re-evaluation of tumor status.

ELIGIBILITY:
Inclusion Criteria:

* Advanced stage,high-risk neuroblastoma
* Histologic proof of neuroblastoma
* Adequate renal function
* ECOG performance status 0-2

Exclusion Criteria:

* Previous therapy

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 1997-10; Primary Completion 2001-04 (Actual); Study Completion 2001-04 (Actual)

PRIMARY OUTCOMES:
Response rate | 5 years

SECONDARY OUTCOMES:
Feasibility/toxicity of an intensification phase of high-dose chemotherapy with topotecan and cyclophosphamide followed by autologous peripheral blood stem cell transplant | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Wayne L. Furman, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Background] Santana VM, Furman WL, Billups CA, Hoffer F, Davidoff AM, Houghton PJ, Stewart CF. Improved response in high-risk neuroblastoma with protracted topotecan administration using a pharmacokinetically guided dosing approach. J Clin Oncol. 2005 Jun 20;23(18):4039-47. doi: 10.1200/JCO.2005.02.097. PMID 15961757
- See also: St. Jude Children's Research Hospital — http://www.stjude.org